CLINICAL TRIAL: NCT04225494
Title: Evaluation of Perioperative Residual Adrenal Function After Extended Multivisceral Resection for Primary Retroperitoneal Soft Tissue Sarcomas: a Prospective Observational Study
Brief Title: Perioperative Residual Adrenal Function After Extended Resection for Retroperitoneal Soft Tissue Sarcomas
Acronym: RAF
Status: Completed | Type: Observational
Sponsor: Fondazione IRCCS Istituto Nazionale dei Tumori, Milano (Other)
Responsible Party: Principal Investigator, Marco Fiore, Principal Investigator, Fondazione IRCCS Istituto Nazionale dei Tumori, Milano
Other Study IDs: 64/19
Record Dates: First submitted 2019-10-01; First posted 2020-01-13 (Actual); Last update posted 2021-10-05 (Actual); Status verified 2021-10

CONDITIONS: Adrenal; Functional Disturbance; Retroperitoneal Sarcoma; Intraoperative Hypotension
Keywords: Retroperitoneal Sarcoma; Surgery; Haemodynamic assessment; Adrenalectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 4 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Early recognition of adrenal function deficit in patients undergoing multivisceral surgery including adrenalectomy for primitive retroperitoneal sarcomas

DETAILED DESCRIPTION:
The extended multivisceral resection of retroperitoneum is the standard treatment for primary retroperitoneal soft tissue sarcomas. This procedure also includes the removal of the healthy adrenal gland ipsilateral to the tumor site.

The investigators think that a such extended surgical approach together with the removal of the adrenal gland may lead to a state of acute adrenal insufficiency and related hemodynamic instability.

In order to recognize this condition the investigators use a low dose ACTH test (Synacthen test) during the 1° and 10° post-operative days.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (age> 18 years)
* Diagnosis of retroperitoneal sarcoma
* Adrenalectomy enbloc included in multivisceral resection
* Voluntary informed written consent

Exclusion Criteria:

* Recurrent and / or metastatic disease
* Patient chronically treated with corticosteroids
* Primary disorders of adrenal gland
* Basal serum cortisol values ≤ 7 µg / dL
* Clinically significant heart disease
* Altered TSH

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary retroperitoneal sarcoma candidated to extended multivisceral resection
Sampling Method: Non-Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2020-08-31 (Actual); Study Completion 2021-05-21 (Actual)

PRIMARY OUTCOMES:
Serum Cortisol peak after low dose Synachten stimulation test. | 1st postoperative day
  Assessment of early postoperative acute adrenal dysfunction.
Serum Cortisol peak after low dose Synachten stimulation test. | 10th postoperative day
  Assessment of postoperative acute adrenal dysfunction.
Serum Cortisol peak after low dose Synachten stimulation test. | 4 months after surgery (only if test positive on 10th postoperative day)
  Assessment of postoperative chronic adrenal dysfunction.

SECONDARY OUTCOMES:
Postoperative morbidity | 30th postoperative day
  Correlation between morbidity according to Clavien-Dindo and postoperative adrenal dysfunction
Vasoactive inotropic score | Intraoperatively and up to 3rd postoperative day
  Correlation between intra- and postoperative usage of vasoactive drugs and postoperative adrenal dysfunction

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione IRCCS Istituto Nazionale dei Tumori, Milan, Lombardy, Italy

IPD SHARING:
Plan to Share IPD: Yes
Individual Participant Data will be shared upon request.
Supporting Information: Study Protocol, ICF, CSR
Time Frame: Five years after study complexion
Access Criteria: Upon motivated request to PI

REFERENCES:
- [Background] Casali PG, Abecassis N, Aro HT, Bauer S, Biagini R, Bielack S, Bonvalot S, Boukovinas I, Bovee JVMG, Brodowicz T, Broto JM, Buonadonna A, De Alava E, Dei Tos AP, Del Muro XG, Dileo P, Eriksson M, Fedenko A, Ferraresi V, Ferrari A, Ferrari S, Frezza AM, Gasperoni S, Gelderblom H, Gil T, Grignani G, Gronchi A, Haas RL, Hassan B, Hohenberger P, Issels R, Joensuu H, Jones RL, Judson I, Jutte P, Kaal S, Kasper B, Kopeckova K, Krakorova DA, Le Cesne A, Lugowska I, Merimsky O, Montemurro M, Pantaleo MA, Piana R, Picci P, Piperno-Neumann S, Pousa AL, Reichardt P, Robinson MH, Rutkowski P, Safwat AA, Schoffski P, Sleijfer S, Stacchiotti S, Sundby Hall K, Unk M, Van Coevorden F, van der Graaf WTA, Whelan J, Wardelmann E, Zaikova O, Blay JY; ESMO Guidelines Committee and EURACAN. Soft tissue and visceral sarcomas: ESMO-EURACAN Clinical Practice Guidelines for diagnosis, treatment and follow-up. Ann Oncol. 2018 Oct 1;29(Suppl 4):iv268-iv269. doi: 10.1093/annonc/mdy321. No abstract available. PMID 30285214
- [Background] Casali PG, Abecassis N, Aro HT, Bauer S, Biagini R, Bielack S, Bonvalot S, Boukovinas I, Bovee JVMG, Brodowicz T, Broto JM, Buonadonna A, De Alava E, Dei Tos AP, Del Muro XG, Dileo P, Eriksson M, Fedenko A, Ferraresi V, Ferrari A, Ferrari S, Frezza AM, Gasperoni S, Gelderblom H, Gil T, Grignani G, Gronchi A, Haas RL, Hassan B, Hohenberger P, Issels R, Joensuu H, Jones RL, Judson I, Jutte P, Kaal S, Kasper B, Kopeckova K, Krakorova DA, Le Cesne A, Lugowska I, Merimsky O, Montemurro M, Pantaleo MA, Piana R, Picci P, Piperno-Neumann S, Pousa AL, Reichardt P, Robinson MH, Rutkowski P, Safwat AA, Schoffski P, Sleijfer S, Stacchiotti S, Sundby Hall K, Unk M, Van Coevorden F, van der Graaf WTA, Whelan J, Wardelmann E, Zaikova O, Blay JY; ESMO Guidelines Committee and EURACAN. Soft tissue and visceral sarcomas: ESMO-EURACAN Clinical Practice Guidelines for diagnosis, treatment and follow-up. Ann Oncol. 2018 Oct 1;29(Suppl 4):iv51-iv67. doi: 10.1093/annonc/mdy096. No abstract available. PMID 29846498
- [Background] Visioni A, Shah R, Gabriel E, Attwood K, Kukar M, Nurkin S. Enhanced Recovery After Surgery for Noncolorectal Surgery?: A Systematic Review and Meta-analysis of Major Abdominal Surgery. Ann Surg. 2018 Jan;267(1):57-65. doi: 10.1097/SLA.0000000000002267. PMID 28437313
- [Background] Trans-Atlantic RPS Working Group. Management of primary retroperitoneal sarcoma (RPS) in the adult: a consensus approach from the Trans-Atlantic RPS Working Group. Ann Surg Oncol. 2015 Jan;22(1):256-63. doi: 10.1245/s10434-014-3965-2. Epub 2014 Oct 15. PMID 25316486
- [Background] Burry L, Little A, Hallett D, Mehta S. Detection of critical illness-related corticosteroid insufficiency using 1 mug adrenocorticotropic hormone test. Shock. 2013 Feb;39(2):144-8. doi: 10.1097/SHK.0b013e31827daf0b. PMID 23324883
- [Background] Annane D, Pastores SM, Rochwerg B, Arlt W, Balk RA, Beishuizen A, Briegel J, Carcillo J, Christ-Crain M, Cooper MS, Marik PE, Umberto Meduri G, Olsen KM, Rodgers SC, Russell JA, Van den Berghe G. Guidelines for the Diagnosis and Management of Critical Illness-Related Corticosteroid Insufficiency (CIRCI) in Critically Ill Patients (Part I): Society of Critical Care Medicine (SCCM) and European Society of Intensive Care Medicine (ESICM) 2017. Crit Care Med. 2017 Dec;45(12):2078-2088. doi: 10.1097/CCM.0000000000002737. PMID 28938253